CLINICAL TRIAL: NCT05941793
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of SNS812 in Participants With Mild to Moderate COVID-19
Brief Title: A Study to Evaluate the Efficacy, Safety, and Concentration of SNS812 in Mild to Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNS812CLCT02
Record Dates: First submitted 2023-07-11; First posted 2023-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mild to Moderate COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): low dosage of IP
  Interventions: Drug: MBS-COV
- Cohort 2 (Experimental): high dosage of IP
  Interventions: Drug: MBS-COV
- Cohort 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBS-COV — MBS-COV for inhalation
  Arms: Cohort 1; Cohort 2
Drug: Placebo — Placebo for inhalation
  Arms: Cohort 3

SUMMARY:
A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of SNS812 in Participants with Mild to Moderate COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults who are 18 and above.
* Body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive).
* Both male and female participants and their partners of childbearing potential must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, tubal sterilization or vasectomy) or must practice complete abstinence from intercourse of reproductive potential from study entry to 3 months after the last day of treatment (excluding women who are not of childbearing potential and men who have been sterilized).
* Participants should be willing to cooperate and able to participate in this study, comply with all protocol requirements, and sign an informed consent.
* Current non-smokers and those who have not smoked within the last 3 months. This includes the use of cigarettes, e-cigarettes, and nicotine replacement products.
* Confirmed SARS-CoV-2 infection as determined by RT-PCR in any specimen collected within 3 days prior to administration.
* Initial onset of signs/symptoms attributable to COVID-19 within 3 days prior to D1 administration and at least 1 of the specified signs/symptoms attributable to COVID-19 present on baseline
* Participants with mild or moderate COVID-19.

Exclusion Criteria:

* Participants who are judged by investigator maybe progressed to severe/critical COVID-19 or need to hospitalization prior to randomization.
* Have SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300 mmHg, respiratory rate ≥30 per minute, heart rate ≥125 per minute
* Participants infected with COVID-19 within 3 months before screening.
* Participants treated with SARS-CoV-2 monoclonal antibodies, antiviral for cure or prevent COVID-19 within 30 days.
* Participants who have received COVID-19 or non-COVID-19 vaccines or human COVID-19 immunoglobulin or convalescent plasma within 3 months before screening, or who plan to receive vaccine (including COVID-19 vaccine booster) during the study.
* Participants who have received systemic or inhaled steroid drugs to cure COVID-19 within 30 days before screening.
* Participants who participate in other clinical trials and use other drugs in the investigation within 1 month or 5 half-life (whichever is longer) before screening.
* Participants with known allergic reactions to the study drug or its excipients.
* The participant has any nasopharyngeal abnormality that may have interfered with nasal absorption, distribution, or study-related evaluations of signs or symptoms
* Participants who have an acute sinusitis, a history of active allergic rhinitis (AR), history of perennial allergic rhinitis (PAR), or current seasonal allergic rhinitis (SAR), or recent viral rhinitis within 2 weeks prior to administration.
* As reported by the participant has severe cardiovascular disease, neurological disease, hematological disease, infectious disease, mental disorder, liver disease, gastrointestinal disease, lung disease, endocrine disease, immune disease or kidney disease, or has a history of the above diseases, or other symptoms known to interfere with the absorption, distribution, metabolism, or excretion of the medicine, or other conditions that the investigator believes will increase the risk of the participant and might interfere with the study conduct and results interpretation.
* Participants who have a history of other malignant tumors within 2 years before enrollment, except for skin basal cell carcinoma, skin squamous cell carcinoma, and carcinoma in situ that have undergone possible curative treatment and have not recurred within 5 years after the start of treatment.
* Participants suspected or diagnosed with active systemic infection, such as bacteria, fungi, viruses or other infections (except COVID-19 infection), or with diseases that the investigator judges will affect the evaluation of the study endpoint.
* Participants who have a known history of hepatitis C virus (HCV), human immunodeficiency virus (HIV), or active HBV infection (if the subject has a history of hepatitis B or has been positive for hepatitis B surface antigen in the past, but the liver function at the baseline period don't meets the exclusion criteria, and the investigator judges that the subject is in a stable period, the subject can be enrolled), or a positive test result for hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at screening.
* Participants with moderate or severe liver disease or kidney disease. And the results of laboratory tests during screening period meet one of the following indicators:

  1. AST or ALT level ≥3 × ULN;
  2. Total bilirubin ≥2 × ULN (≥3 × ULN for Gilbert's syndrome);
  3. Total WBC 2,500/mm3 or absolute neutrophil count <1500/mm3.
  4. eGFR < 30 mL/min, calculated by CKD-EPI formula.
  5. Platelet count < 80,000/mm3
* Ventilatory dysfunction or inability to use a nebulizer with a face mask.
* Females who are pregnant or breastfeeding.
* Any other situation that, judged by the investigator, may affect the subject to provide informed consent or to comply with the study protocol, or may affect the study results or their own safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events,and Serious Adverse Events (SAEs) | 2 months

SECONDARY OUTCOMES:
Time (days) to sustained alleviation of all targeted signs/symptoms through Day 28. | 28 days
Time (days) to sustained resolution of all targeted signs/symptoms through Day 28 | 28 days
Proportion of participants with sustained alleviation of all targeted signs/symptoms through Day 60. | 60 days
Proportion of participants with sustained resolution of all targeted signs/symptoms through Day 60. | 60 days
Time (days) to sustained alleviation of Shortness of breath through Day 28. | 28 days
Time (days) to sustained resolution of Shortness of breath through Day 28. | 28 days
Time (days) to sustained alleviation of each sign/symptom through Day 28. | 28 days
Time (days) to sustained resolution of each sign/symptom through Day 28. | 28 days
Proportion of participants with sustained alleviation of each sign/symptom through Day 60. | 60 days
Proportion of participants with sustained resolution of each sign/symptom through Day 60. | 60 days

CONTACTS AND LOCATIONS:
Locations (5):
- Velocity Clinical Research, Salt Lake City, Utah, United States
- Taiwan (4):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei